CLINICAL TRIAL: NCT04970407
Title: A Phase I, Randomised, Double-blind, Parallel-group, Single-centre Comparative Study to Evaluate the Pharmacodynamic Profile of Dysport®, Botox®, and Xeomin® in the Extensor Digitorum Brevis (EDB) Model in Healthy Adult Male Participants
Brief Title: A Comparative Study to Evaluate the Effects and Mechanism of Action of Dysport®, Botox® and Xeomin® in the Extensor Digitorum Brevis Model in Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D-FR-52120-279; 2021-000802-14 (EudraCT Number)
Record Dates: First submitted 2021-07-02; First posted 2021-07-21 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA; incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dysport® (Experimental): 40 Units (U) Intramuscular (IM) injection at day 1.
  Interventions: Biological: Botulinum toxin type A
- Botox® (Active Comparator): 16U IM at day 1.
  Interventions: Biological: Botulinum toxin type A
- Xeomin® (Active Comparator): 16U IM at day 1.
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A — Intramuscular Injection, concentration 300 units (U)
  Other Names: abobotulinumtoxinA (Dysport®)
  Arms: Dysport®
Biological: Botulinum toxin type A — Intramuscular Injection, concentration 50 U
  Other Names: onabotulinumtoxinA (Botox®)
  Arms: Botox®
Biological: Botulinum toxin type A — Intramuscular Injection, concentration 50 U
  Other Names: incobotulinumtoxinA (Xeomin®)
  Arms: Xeomin®

SUMMARY:
Study aimed at comparing the pharmacodynamic profile (including duration of action) of three commercialized toxins by measuring the action potential of the injected muscle (extensor digitorum brevis)

ELIGIBILITY:
Inclusion Criteria:

* Participant must be between18 to 65 years of age inclusive, at the time of signing the informed consent
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs and cardiac monitoring
* A body mass index (BMI) within the range 18 and 30 kg/m2 (inclusive).

Exclusion Criteria:

* Any medical condition that may put the participant at risk with exposure to BoNT, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disease that might interfere with neuromuscular function
* Previous treatment with botulinum toxin (BoNT) (any serotype) during the past 6 months
* Known hypersensitivity to any of the components of the Dysport/ Botox/ Xeomin formulation (which includes human serum albumin, lactose, sucrose) or allergy to cow's milk protein
* Use of agents that could interfere with neuromuscular transmission, including calcium channel blockers, penicillamine, aminoglycosides, lincosamides, polymixins, magnesium sulphate, anticholinesterases, succinylcholine and quinidine

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Mac Research Clinical research Unit, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2023/09/08121839/Study-D-FR-52120-279-Dysport-lay-summary.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase I, randomized, double-blind study was conducted in healthy adult male participants at a single investigational site in United Kingdom between 06 Jul 2021 and 08 Jun 2022. The purpose of this study was to compare the duration of action on compound muscle action potential (CMAP) of the extensor digitorum brevis (EDB) muscle injected with either Dysport 40 units (U), Botox 16 U or Xeomin 16 U.
Pre-assignment Details: This study consisted of a 14-day screening period, a double-blind period including treatment administration on Day 1, and follow-up period up to 40 weeks. A total of 45 male participants were randomized in a 1:1:1 ratio to receive treatment with Dysport 40 U, Botox 16 U or Xeomin 16 U respectively.
Groups:
- Dysport 40 U: Participants received a single intramuscular (IM) injection of Dysport 40 U in the EDB muscle on Day 1.
- Botox 16 U: Participants received a single IM injection of Botox 16 U in the EDB muscle on Day 1.
- Xeomin 16 U: Participants received a single IM injection of Xeomin 16 U in the EDB muscle on Day 1.
Period: Overall Study
Arm/Group | Dysport 40 U | Botox 16 U | Xeomin 16 U
Started | 15 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Randomized set consisted of all participants who were randomized to study treatment. A participant was considered as randomized if a study intervention group was randomly assigned.
Groups:
- Dysport 40 U: Participants received a single IM injection of Dysport 40 U in the EDB muscle on Day 1.
- Total: Total of all reporting groups
Arm/Group | Dysport 40 U | Botox 16 U | Xeomin 16 U | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (11.3) | 35.3 (12.3) | 34.8 (13.9) | 35.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 15 | 15 | 15 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Adjusted Mean (AM) Percentage (%) of CMAP Total Amplitude at Week 28
Description: The CMAP procedure was performed on the injected foot by a neurophysiologist. Percentage relative to baseline was calculated as (value at Week 28 [mean of the 3 measurements]/baseline value) multiplied by (*) 100. The adjusted mean was obtained from a mixed-effects model for repeated measures (MMRM) model with Fisher scoring. Baseline was defined as the last non-missing measurement taken prior to study drug administration. Baseline value used for this analysis was the average of 6 measurements, the 3 measurements at screening and the 3 measurements at baseline.
Time Frame: Baseline (Day 1) and Week 28
Population: The Pharmacodynamic (PD) analysis set consisted of all participants from the randomized set who received the appropriate dose of study treatment and had CMAP recorded for baseline and at least 1 post-baseline assessment.
Measure: Mean (Standard Error); unit: % of AM of CMAP total amplitude
Arm/Group | Dysport 40 U | Botox 16 U | Xeomin 16 U
Number analyzed (Participants) | 15 | 15 | 15
% of AM of CMAP total amplitude | 73.62 (5.26) | 74.78 (5.26) | 84.23 (5.25)
Statistical Analysis 1: Comparison: Dysport 40 U vs Botox 16 U; The adjusted mean, standard error (SE) and 95% confidence interval (CI) of the adjusted mean as well as difference in % relative to baseline and p-value were obtained from a MMRM with Fisher scoring with treatment, time (corresponding to all study visits when CMAP was measured), treatment by time interaction and baseline CMAP amplitude as factors and an unstructured variance covariance matrix; Test type: Superiority; p = 0.8769, MMRM model; Treatment difference = -1.16, 95% CI 2-sided [-16.25 to 13.93]
Statistical Analysis 2: Comparison: Dysport 40 U vs Xeomin 16 U; The adjusted mean, SE and 95% CI of the adjusted mean as well as difference in % relative to baseline and p-value were obtained from a MMRM with Fisher scoring with treatment, time (corresponding to all study visits when CMAP was measured), treatment by time interaction and baseline CMAP amplitude as factors and an unstructured variance covariance matrix; Test type: Superiority; p = 0.1620, MMRM model; Treatment difference = -10.61, 95% CI 2-sided [-25.69 to 4.47]

2. Secondary Outcome: Change From Baseline in AM % of CMAP Total Amplitude at Week 40
Description: The CMAP procedure was performed on the injected foot by a neurophysiologist. It was measured as percentage relative to baseline defined as CMAP at the corresponding visit (mean of the 3 measurements)/CMAP at baseline (mean of the 6 measurements)*100. The adjusted mean was obtained from a MMRM model with Fisher scoring. Baseline was defined as the last non-missing measurement taken prior to study drug administration. Baseline value used for this analysis was the average of 6 measurements, the 3 measurements at screening and the 3 measurements at baseline.
Time Frame: Baseline (Day 1) and Week 40
Population: The PD analysis set consisted of all participants from the randomized set who received the appropriate dose of study treatment and had CMAP recorded for baseline and at least 1 post-baseline assessment.
Measure: Mean (Standard Error); unit: % of AM of CMAP total amplitude
Arm/Group | Dysport 40 U | Botox 16 U | Xeomin 16 U
Number analyzed (Participants) | 15 | 15 | 15
% of AM of CMAP total amplitude | 77.10 (5.09) | 81.83 (5.10) | 92.01 (5.09)

3. Secondary Outcome: Percentage of Participants With Recovery of CMAP Total Amplitude
Description: The recovery was considered to be reached for all the visits occurring after the time to recovery, that is (i.e.) the first visit for which CMAP total amplitude returned to at least 85% of the baseline value. Percentage of participants with recovery of CMAP total amplitude was analyzed at Weeks 28 and 40.
Time Frame: At Weeks 28 and 40
Population: The PD analysis set consisted of all participants from the randomized set who received the appropriate dose of study treatment and had CMAP recorded for baseline and at least 1 post-baseline assessment. Only those participants who showed recovery at Weeks 28 and 40 were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dysport 40 U | Botox 16 U | Xeomin 16 U
Number analyzed (Participants) | 15 | 15 | 15
percentage of participants
  Week 28 | 33.3 [11.8 to 61.6] | 26.7 [7.8 to 55.1] | 53.3 [26.6 to 78.7]
  Week 40 | 33.3 [11.8 to 61.6] | 33.3 [11.8 to 61.6] | 66.7 [38.4 to 88.2]

4. Secondary Outcome: Time to Onset of Action of Study Intervention
Description: Time to onset of action was defined as the first timepoint when EDB CMAP total amplitude was less or equal to 85% of the baseline value.
Time Frame: From Baseline (Day 1) up to Week 40
Population: as for outcome 2
Measure: Median (Full Range); unit: weeks
Arm/Group | Dysport 40 U | Botox 16 U | Xeomin 16 U
Number analyzed (Participants) | 15 | 15 | 15
weeks | 1.00 [0.7 to 1.6] | 1.00 [0.7 to 1.1] | 1.00 [0.9 to 4.0]

5. Secondary Outcome: Duration of Response
Description: Duration of response was calculated as time to recovery of CMAP total amplitude - time to onset. Time to recovery was defined as the first timepoint where EDB CMAP total amplitude returned to at least 85% of the baseline value.
Time Frame: From Baseline (Day 1) up to Week 40
Population: The PD analysis set consisted of all participants from the randomized set who received the appropriate dose of study treatment and had CMAP recorded for baseline and at least 1 post-baseline assessment. Only those participants who showed recovery before the end of the study were analyzed.
Measure: Median (Full Range); unit: weeks
Arm/Group | Dysport 40 U | Botox 16 U | Xeomin 16 U
Number analyzed (Participants) | 5 | 5 | 10
weeks | 18.29 [7.0 to 19.0] | 10.86 [7.3 to 31.4] | 17.07 [3.1 to 38.6]

6. Secondary Outcome: Percentage of Maximal Inhibition (Maximal Effect) of CMAP Total Amplitude
Description: Maximal inhibition was defined as the maximal measured inhibition of CMAP total amplitude of stimulated EDB.
Time Frame: Up to Week 40
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of inhibition
Arm/Group | Dysport 40 U | Botox 16 U | Xeomin 16 U
Number analyzed (Participants) | 15 | 15 | 15
percentage of inhibition | 39.79 [31.23 to 48.35] | 38.55 [33.99 to 43.10] | 44.99 [36.68 to 53.30]

7. Secondary Outcome: Number of Participants Who Achieved Maximal Effect of CMAP Total Amplitude
Description: Time to maximal effect was defined on an individual basis as the time between baseline and the timepoint of maximal inhibition of CMAP amplitude of stimulated EDB. Participants with maximal effect of CMAP total amplitude were reported.
Time Frame: At Weeks 1, 4, 8 and 20
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dysport 40 U | Botox 16 U | Xeomin 16 U
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Week 1 | 11 | 13 | 11
  Week 4 | 2 | 1 | 4
  Week 8 | 1 | 1 | 0
  Week 20 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the study drug administration (Day 1) up to Week 40
Description: The Safety analysis set consisted of all participants who received at least 1 dose of study treatment.
Arm/Group | Dysport 40 U | Botox 16 U | Xeomin 16 U
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 10/15 | 2/15 | 5/15
Other Adverse Events (participants affected / at risk) | 11/15 | 10/15 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport 40 U (N=15) | Botox 16 U (N=15) | Xeomin 16 U (N=15)
Covid-19 (Infections and infestations) | 10 (10) | 2 (2) | 4 (4)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport 40 U (N=15) | Botox 16 U (N=15) | Xeomin 16 U (N=15)
Viral infection (Infections and infestations) | 2 (2) | 2 (3) | 4 (4)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 5 (7)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT04970407/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT04970407/SAP_001.pdf